CLINICAL TRIAL: NCT04623684
Title: Efficacy and Safety of Mydriatic Microdrops Compared With Standard Drops for Retinopathy of Prematurity (ROP) Screening: a Pilot Randomized Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Asimina Mataftsi, Associate Professor in Ophthalmology, Paediatric Ophthalmology and Strabismus, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: 170/10-03-2020
Record Dates: First submitted 2020-10-31; First posted 2020-11-10 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Retinopathy of Prematurity
Keywords: microdrops; mydriasis; dilating drops; retinopathy of prematurity; ROP; screening
MeSH Terms: conditions — Retinopathy of Prematurity; Mydriasis | interventions — Phenylephrine; Tropicamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Mydriasis with microdrops
  Interventions: Drug: Microdrop administration [phenylephrine 1.67% + tropicamide 0.33% (drop volume: 6-7 μL)]
- Control Group (Active Comparator): Mydriasis with standard drops
  Interventions: Drug: Standard drop administration [phenylephrine 1.67% + tropicamide 0.33% (drop volume: 28-34 μL)]

INTERVENTIONS:
Drug: Microdrop administration [phenylephrine 1.67% + tropicamide 0.33% (drop volume: 6-7 μL)] — 1 drop (6-7 μL) for 3 doses, 5 minutes' intervals
  Arms: Study Group
Drug: Standard drop administration [phenylephrine 1.67% + tropicamide 0.33% (drop volume: 28-34 μL)] — 1 drop (28-34 μL) for 3 doses, 5 minutes' intervals
  Arms: Control Group

SUMMARY:
The purpose is to assess whether the use of microdrop instillation of phenylephrine 1.67% and tropicamide 0.33% maintains mydriatic efficacy while presents an improved safety profile compared with standard drops of phenylephrine 1.67% and tropicamide 0.33%, which is routine care for pupil dilation during retinopathy of prematurity (ROP) screening in our neonatal intensive care unit.

DETAILED DESCRIPTION:
A pilot prospective randomized crossover clinical trial is conducted for assessing the mydriatic efficacy and safety of microdrops (6-7 μL) compared with standard drops (28-34 μL) for retinopathy of prematurity screening. A random number table was used to allocate participants into either a) receiving standard drop on their first and microdrop on their second screening examination a week later, or b) receiving microdrop first and standard drop a week later. The mydriatic agent contains phenylephrine 1.67% and tropicamide 0.33%, which derives from compounding the commercial phenylephrine 5% with the commercial tropicamide 0.5% in volume ratio 1:2.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants undergoing screening for ROP, i.e.

* with gestational age (GA) < 32 weeks and/or birth weight (BW) < 1501 grams
* infants of greater GA and BW with increased comorbidity, e.g. sepsis, prolonged need for oxygen supplementation etc.

Exclusion Criteria:

* Unstable clinical condition
* Suspicion of cardiovascular disease
* Severe congenital anomalies
* Clinical syndromes
* Traumatic apoptosis of the corneal epithelium
* Corneal ulcer
* Anatomical variations of the anterior segment

Ages: 30 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Mydriatic efficacy: mm of pupil diameter (left and right eye) | 45 minutes after the first drop instillation
Mydriatic efficacy: mm of pupil diameter (left and right eye) | 90 minutes after the first drop instillation

SECONDARY OUTCOMES:
Mydriatic efficacy: mm of pupil diameter (left and right eye) | 120 minutes after the first drop instillation
Systemic side effects: measurements of Heart Rate (bpm) | 45 minutes after the first drop instillation
Systemic side effects: measurements of Heart Rate (bpm) | 90 minutes after the first drop instillation
Systemic side effects: measurements of Heart Rate (bpm) | 120 minutes after the first drop instillation
Systemic side effects: measurements of oxygen saturation (SpO2) (%) | 45 minutes after the first drop instillation
Systemic side effects: measurements of oxygen saturation (SpO2) (%) | 90 minutes after the first drop instillation
Systemic side effects: measurements of oxygen saturation (SpO2) (%) | 120 minutes after the first drop instillation
Systemic side effects: measurements of Blood Pressure (Systolic, Diastolic and Mean Blood Pressure) (mmHg) | 45 minutes after the first drop instillation
Systemic side effects: measurements of Blood Pressure (Systolic, Diastolic and Mean Blood Pressure) (mmHg) | 90 minutes after the first drop instillation
Systemic side effects: measurements of Blood Pressure (Systolic, Diastolic and Mean Blood Pressure) (mmHg) | 120 minutes after the first drop instillation
Systemic side effects: measurements of Blood Pressure (Systolic, Diastolic and Mean Blood Pressure) (mmHg) | Hourly for the first 24 hours after mydriasis
Local side effects: periorbital pallor, eyelid swelling, flushing | 45 minutes after the first drop instillation
Adverse events including apnea, increased gastric residuals, inhibited duodenal motor activity, delayed gastric emptying, feeding intolerance, abdominal distension, vomiting, paralytic ileus, acute gastric dilatation and necrotizing enterocolitis (NEC) | During the 24 hours after mydriasis for ROP screening
Number of participants with non-adequate mydriasis to fully visualize peripheral fundus according to the examiner | Upon eye examination (45 to 90 minutes after the first drop)

CONTACTS AND LOCATIONS:
Locations (1):
- "Papageorgiou" General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lynch MG, Brown RH, Goode SM, Schoenwald RD, Chien DS. Reduction of phenylephrine drop size in infants achieves equal dilation with decreased systemic absorption. Arch Ophthalmol. 1987 Oct;105(10):1364-5. doi: 10.1001/archopht.1987.01060100066027. PMID 3662909
- [Background] Elibol O, Alcelik T, Yuksel N, Caglar Y. The influence of drop size of cyclopentolate, phenylephrine and tropicamide on pupil dilatation and systemic side effects in infants. Acta Ophthalmol Scand. 1997 Apr;75(2):178-80. doi: 10.1111/j.1600-0420.1997.tb00119.x. PMID 9197568
- [Background] Seliniotaki AK, Prousali E, Lithoxopoulou M, Kokkali S, Ziakas N, Soubasi V, Mataftsi A. Alternative mydriasis techniques for retinopathy of prematurity screening. Int Ophthalmol. 2020 Dec;40(12):3613-3619. doi: 10.1007/s10792-020-01542-x. Epub 2020 Aug 9. PMID 32772218
- [Result] Seliniotaki AK, Lithoxopoulou M, Talimtzi P, Georgiou E, Diamanti E, Ziakas N, Haidich AB, Mataftsi A. Efficacy and safety of mydriatic microdrops for retinopathy of prematurity screening: an external pilot crossover randomized controlled trial. J Perinatol. 2022 Mar;42(3):371-377. doi: 10.1038/s41372-021-01229-w. Epub 2021 Oct 15. PMID 34654903